CLINICAL TRIAL: NCT04565405
Title: Microbiological Evaluation of the Efficacy of Water to Clean Tracheostomy Inner Cannulas: A Randomized Control Trial
Brief Title: Microbiological Evaluation of the Efficacy of Water to Clean Tracheostomy Inner Cannulas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Chan Hong Eng, Senior Nurse Clinician, Changi General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Inner Cannula
Record Dates: First submitted 2020-09-08; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Tracheostomy Complication
Keywords: Tracheostomy; Inner cannulas; Decontamination; Microbiological evaluation
MeSH Terms: interventions — Detergents

STUDY DESIGN:
Intervention Model Description: This is a single centre, single blinded, randomized cross over study comparing two decontamination procedures Detergent (A) and Sterile water (B) on inner cannulas.
  To avoid the influence of confounding covariates, we propose to have a cross over study. The cross over patient will act as his own control. The selected patients will be randomly allocated to sequence AB or BA in 1:1 fashion using permuted blocks with different block sizes.
  The change of sequence A > B and B > A will take place only after minimum of 24 hours after the first part of sequence has been completed.
Who Masked: Participant, Outcomes Assessor
Masking Description: Eligible patients will be randomized in 1:1 fashion using permuted blocks with different block sizes. The subjects and lab operators will be blinded to the block size and randomization. In the event unmasking need to be performed, a staff who is not involved in this study from Clinical Trial Unit will perform the unmasking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB (Detergent (A) followed by sterile water (B)) (Experimental): Sequence: Detergent (A) followed by sterile water (B)
  The inner cannula will be cleaned with commercially available tracheostomy cleaning fluid / powder (Ex: Trachoe - Kapitex healthcare, UK) in the first visit, and then cleaned with sterile water in the second visit, at a minimum period of 24 hrs apart. Laboratory analysis of colony counts will be conducted on the saline flushing pre- and post-decontamination for each washing.
  Interventions: Other: Detergent; Other: Sterile water
- BA (Sterile water (B) followed by detergent (A)) (Experimental): Sequence: Sterile water (B) followed by detergent (A)
  The inner cannula will be cleaned with sterile water in the first visit, and then cleaned with commercially available tracheostomy cleaning fluid / powder (Ex: Trachoe - Kapitex healthcare, UK) in the second visit, at a minimum period of 24 hrs apart. Laboratory analysis of colony counts will be conducted on the saline flushing pre- and post-decontamination for each washing.
  Interventions: Other: Detergent; Other: Sterile water

INTERVENTIONS:
Other: Detergent — The tracheostomy inner cannulas will be washed with detergent.
Other: Sterile water — The tracheostomy inner cannulas will be washed with sterile water.

SUMMARY:
Biofilms pose a potential risk with reusable inner cannulas, by increasing the risk of infection. Effective decontamination is vital in eliminating these biofilms. An appropriate method of cleaning and decontamination to make inner cannula safe for reuse should be practiced. The current recommendations for cleaning inner cannula are varied with multiple techniques being put forth. The current practice of using sterile water to clean inner cannula is not supported by strong evidence. This Randomized Controlled Study looks into the microbiological efficacy of sterile water in cleaning inner cannulas.

DETAILED DESCRIPTION:
Tracheostomy Care of Patients:

The tracheostomy care of all patients included in the study will be the same as any other tracheostomy patient in the hospital, as directed by the tracheostomy care nursing policy. Before study procedure, inner cannula is to be checked to ensure it is not clogged with secretion, any secretion is to be removed with suction.

Decontamination methods:

Patients may fall under group A or group B as determined by the random allocation.

Patients in decontamination group A: Detergent

Pre Decontamination:

* The inner cannula care will be removed using aseptic precautions.
* 10 ml of normal saline will be flushed along the inner surface in an uniform manner over 30 seconds. The inner cannula will be turned gently to ensure that the entire inner surface has been flushed by Normal Saline.
* The solution will be collected in the sterile bottle and sent for laboratory analysis of colony counts.
* Small proportion of pre decontamination samples will be randomly selected for typing and naming of organisms.

Decontamination:

* Inner cannula will be cleaned with commercially available tracheostomy cleaning fluid / powder (Ex: Trachoe - Kapitex healthcare, UK).
* The cleaning is done as per manufacturers recommendation.

Post Decontamination:

* Using aseptic technique, 10 ml of normal saline will be flushed along the inner surface in an uniform manner over 30 seconds. The inner cannula will be turned gently to ensure that the entire inner surface has been flushed by Normal Saline.
* The solution will be collected in the sterile bottle and sent for laboratory analysis of colony counts.

Patients in decontamination group B: Water

Pre Decontamination:

* The inner cannula care will be removed using aseptic precautions.
* 10 ml of normal saline will be flushed along the inner surface in an uniform manner over 30 seconds. The inner cannula will be turned gently to ensure that the entire inner surface has been flushed by Normal Saline.
* The solution will be collected in the sterile bottle and sent for laboratory analysis of colony counts.
* Small proportion of pre decontamination samples will be randomly selected for typing and naming of organisms.

Decontamination:

• Inner cannula is cleaned as per the current tracheostomy care guidelines as directed by the Nursing Policy for Tracheostomy Care, Changi General Hospital. Only Sterile water is recommended as per the policy.

Post Decontamination:

* Using aseptic technique, 10 ml of normal saline will be flushed along the inner surface in an uniform manner over 30 seconds. The inner cannula will be turned gently to ensure that the entire inner surface has been flushed by Normal Saline.
* The solution will be collected in the sterile bottle and sent for laboratory analysis of colony counts.

Crossover of Patients:

To avoid the influence of confounding covariates, we propose to have a cross over study. The cross over patient will act as his own control. The selected patients will be randomly allocated to sequence AB or BA in 1:1 fashion using permuted blocks with different block sizes. The subjects and lab operators will be blinded to the block size and randomization.

The change of sequence A > B and B > A will take place only after minimum of 24 hours after the first part of sequence has been completed. Exclusion criteria will still be applicable after completion of one part of the sequence. Small proportion of pre decontamination samples will be randomly selected for typing and naming of organisms.

Lab Method for Colony Counts:

From the flush solution, 100 microlitres and further sequential serial dilutions of 1:10 (in saline) are cultured directly onto blood agar plates. After 72 hours aerobic incubation at 35oC, all plates are examined and growth from plates with 10 to 100 colonies per plate are counted. Total bacterial growth will be expressed as colony-forming unit (cfu)/ml.

Small proportion of pre decontamination samples will be randomly selected for typing and naming of organisms.

ELIGIBILITY:
Inclusion Criteria:

* All patients under the purview of the tracheostomy care team at Changi General Hospital will be considered for inclusion in the study.
* Patients aged between 21 - 100 years
* Patients with a tracheostomy tube in situ

Exclusion Criteria:

* Pregnant women
* Prisoners
* Patients with documented HIV, Hep C, Hep B
* Patients with active tuberculosis
* Patients being treated in Intensive Care Units
* Patients with ongoing antibiotic treatment or within the last 24 hours
* Unstable patients needing cardiorespiratory support

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-11-16 (Estimated); Study Completion 2020-11-16 (Estimated)

PRIMARY OUTCOMES:
Efficacy of water vs detergent in cleaning tracheostomy inner cannulas | 1 week
  Compare the colony forming units / ml before and after cleaning with water vs detergent

SECONDARY OUTCOMES:
Economic evaluation | 2 years
  Compare the expenses incurred from cleaning the inner cannulas using water vs detergent
Microbiological evaluation | 2 weeks
  Compare the profile of bacteria identified from a proportion of samples sent for bacterial culture between the water and detergent groups

CONTACTS AND LOCATIONS:
Overall Officials: Hong Eng Chan, Principal Investigator — Changi General Hospital
Locations (1):
- Clinical Trials & Research Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorling G, Belin AL, Hellstrom C, Schedin U, Ransjo U, Alenius M, Johansson UB. Tracheostomy inner cannula care: a randomized crossover study of two decontamination procedures. Am J Infect Control. 2007 Nov;35(9):600-5. doi: 10.1016/j.ajic.2006.11.006. PMID 17980239